CLINICAL TRIAL: NCT04088968
Title: STRONG for Surgery & Strong for Life - Against All Odds: Intensive Prehabilitation Including Smoking, Nutrition, Alcohol and Physical Activity for Risk Reduction in Cancer Surgery
Brief Title: STRONG for Surgery & Strong for Life - Against All Odds: Intensive Prehabilitation for Risk Reduction in Cancer Surgery
Acronym: STRONG-CS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Hanne Tonnesen, Professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STRONG Cancer Surg (COMPAS)
Record Dates: First submitted 2019-07-08; First posted 2019-09-13 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Risk Reduction; Urological Cancer; Surgery; Life Style
Keywords: Postoperative complications; Prehabilitation; Surgical risk reduction; Smoking; Alcohol drinking; Physical activity; Malnutrition; Obesity; Patient preferences; Randomised controlled trial
MeSH Terms: conditions — Risk Reduction Behavior; Urologic Neoplasms; Postoperative Complications; Smoking; Alcohol Drinking; Motor Activity; Malnutrition; Obesity; Patient Preference | interventions — Preoperative Exercise; Ethanol; Exercise; Nutritional Support; Adiposity

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trials, Implementation feasibilty trial, Interviews nested
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will not know if patients were allocated to intervention or control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Experimental): Intervention: Patients allocated to the intervention group receive weekly counselling sessions in 6 weeks as an integrated prehabilitation program tailored to meet the individual patient's need for risk reduction at surgery. It is introduced via the surgical 'Engage in the process of change'. The smoking and alcohol cessation intervention follows the Gold Standard Programme and patients in the intervention group are introduced to a standardized exercise training programme taking individualized needs into account. Nutritional support is also individualized.
  Interventions: Behavioral: Prehabilitation
- Treatment as usual (No Intervention): Treatment as ususal covers shorter interventions, e.g. advice, brief counselling, and handing out the national folders on smoking and alcohol and surgery. Patients are ensured that they are free to access support to lifestyle changes in the community.

INTERVENTIONS:
Behavioral: Prehabilitation — Patients screened positive for minimun 1 SNAP factor will be offered enrollment in the study and have an individualized plan for the prehabilitation intervention.
  Other Names: smoking cessation, alcohol cessation, physical activity, nutritional support for malnutrition and obesity
  Arms: Prehabilitation

SUMMARY:
Despite knowledge about the effect of preventive measures in lifestyle, smoking,nutrition, alcohol and physical activity (SNAP), there is a lack of systematic assessment of the overall lifestyle of the patient before surgery and knowledge about how lifestyle interventions can be organized in connection with cancer surgery. The intention with prehabilitation is to optimize the individual's risk factors and personal burdens that can affect the clinical and patient reported outcomes after surgery. The aim of this study is to evaluate the efficacy of intensive SNAP interventions compared to treatment as usual (TAU) in ptt undergoing urological cancer surgery on surgical risk reduction.

DETAILED DESCRIPTION:
The project contains three clinical intervention studies, in total including 100 urological cancer patients screened positive for at least 1 SNAP factor:

I. Efficacy and preferences of intensive SNAP-Interventions among patients with at least one SNAP factor and undertaking neo-adjuvant chemotherapy before radical cystectomy. A randomised controlled trial with nested interviews (42 patients).

II. Implementation and preferences of intensive SNAP-Interventions among patients with kidney cancer undergoing nephrectomy/partial nephrectomy. An implementation feasibility study including interviews (20 patients).

III. Reach out and effect as well as preferences of perioperative intensive smoking cessation intervention via the municipality clinic compared to the surgical department among smokers with non-invasive bladder cancer treated with Trans-Urethral Resection of the Bladder (TUR-B). A randomised controlled trial with nested interviews (38 patients).

The intervention groups receive minimum five educational sessions tailored to individual needs over six weeks perioperatively. The control groups receive standard care.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years scheduled for cystectomy due to bladder cancer
* Referral to neoadjuvant chemotherapy
* Screened positive for minimum 1 SNAP factor
* Signed informed consent

Exclusion Criteria:

* Pregnancy and breastfeeding
* Allergy to pharmaceutical support (Nicotine Replacement Therapy, Disulfiram)
* Contraindications to exercise.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with risk reduction at surgery | End of intervention/ at surgery
  Corresponding at least 1 step for 1 or more risky lifestyles (but only smoking in study III) on the ASA-score (American Society of Anaesthesiologists physical status classification from 1-5, lower is better)

SECONDARY OUTCOMES:
Health related quality of life (HRQoL) | 6 weeks/day at surgery, at 1 month and through study completion, an average of 6 months
  Mean difference of HRQoL between groups measured with EQ5D (5 level quality of life score (level 1 =no problems, level 2-5 =problems)
Number of patients with any postoperative complication | 30 days
  Scored by the Comprehensive Complication Index, a linear scale ranging from 0 (no complication) to 100 (death)
Number of successful tobacco quitters | 6 weeks/day at surgery, at 1 month and through study completion, an average of 6 months
  Successful quitting smoking: Study I+ II+ III
  * Successful quitting alcohol intake at 6 weeks and below risky limits at 6 months: Study I.
  * Physical activity at least 30 minutes per day: Study I.
  * Malnutrition: Not at risk of malnutrition: Study I. Obesity: 5% -10 % loss of body fat mass and below 1% gain of body fat mass at 6 months (without developing malnutrition)
Number of successful alcohol quitters | 6 weeks/day at surgery, at 1 month and through study completion, an average of 6 months
  Successful quitting alcohol: Study I+II
Number of patients being physical active at least 30 min per day | 6 weeks/day at surgery, at 1 month and through study completion, an average of 6 months
  Minutes physical active measured by an accelerometer (longer time is better) : Study I+II
Number of patients not at risk of malnutrition | 6 weeks/day at surgery, at 1 month and through study completion, an average of 6 months
  NRS2002 (Nutritional Risk Screening 2002) score>2. Lower is better: Study I+II
Number of patients not at risk of obesity | 6 weeks/day at surgery, at 1 month and through study completion, an average of 6 months
  BMI (Body Mass Index)<30. Lower is better : Study I+II
Number of patients with improved frailty level | 6 weeks/day at surgery, at 1 month and through study completion, an average of 6 months
  Measured by Lammers definition: Lower is better: Study I+II+III
Number of patients with any reduction in lifestyle | 6 weeks/day at surgery, at 1 month and through study completion, an average of 6 months
  Measured by yes/no. Study I+II+III

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Tonnesen, Professor MD, Principal Investigator — WHOCC, The Parker Institute, Bispebjerg-Frederiksberg Hospital, RegH, Copenhagen
Locations (1):
- Dept Urology 2112, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Region H, Denmark

REFERENCES:
- [Derived] Tonnesen H, Lydom LN, Joensen UN, Egerod I, Pappot H, Lauridsen SV. STRONG for Surgery & Strong for Life - against all odds: intensive prehabilitation including smoking, nutrition, alcohol and physical activity for risk reduction in cancer surgery - a protocol for an RCT with nested interview study (STRONG-Cancer). Trials. 2022 Apr 21;23(1):333. doi: 10.1186/s13063-022-06272-2. PMID 35449008